CLINICAL TRIAL: NCT07148843
Title: Cannabidiol as an Adjunct Treatment for Alcohol Withdrawal and Craving
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00519608
Record Dates: First submitted 2025-08-19; First posted 2025-08-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder (AUD); Withdrawal From Addictive Substance; Detoxification; Craving
Keywords: alcohol abstinence; alcohol withdrawal treatment; detoxification
MeSH Terms: conditions — Alcoholism; Alcohol Abstinence | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, the study team, CRU medical staff, and statistician assessing outcomes will be blinded to the study. The pharmacists will randomize subjects to study arms and if needed can reveal intervention if needed (e.g., clinical care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 10 mg/kg CBD (Active Comparator): low dose CBD
  Interventions: Drug: Cannabidiol (CBD)
- 20 mg/kg CBD (Active Comparator): high dose CBD
  Interventions: Drug: Cannabidiol (CBD)
- placebo (Placebo Comparator): Placebo (no CBD)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol (CBD) — Cannabidiol
  Arms: 10 mg/kg CBD; 20 mg/kg CBD
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
Cannabidiol (CBD), one of the most prevalent cannabinoids in cannabis (marijuana) has been shown to reduce alcohol withdrawal symptoms in laboratory animals. In people without alcohol use disorder (AUD), CBD has been show to be effective in reducing anxiety, sleep problems, and seizures; all of these are common symptoms of alcohol withdrawal. This randomized placebo-controlled clinical trial will evaluate the potential of CBD to improve alcohol withdrawal symptoms and reduce craving during acute abstinence among individuals with moderate-to-severe AUD. Adult participants with moderate-to-severe AUD will be admitted to an inpatient research unit at the Johns Hopkins Hospital for a 5-day, 4-night stay that includes alcohol abstinence with management of their alcohol withdrawal. In addition to standard care, participants will receive CBD or placebo (no CBD), complete assessments of withdrawal, sleep quality and provide breath and blood samples.

DETAILED DESCRIPTION:
Alcohol withdrawal during acute abstinence represents a major health threat to millions of individuals struggling with alcohol use disorder (AUD): it has been associated with complications in patients admitted for medically supervised withdrawal including seizures and delirium tremens (the latter of which can be fatal if not managed appropriately) and can interfere with treatment efforts. Benzodiazepines, such as lorazepam (Ativan) represent the first-line treatments for control of alcohol withdrawal, yet higher doses of benzodiazepines required to manage more complicated withdrawal cases increase risk of respiratory depression and delirium. Furthermore, a growing frequency of benzodiazepine shortages (at least 20 shortages within the previous ten years lasting a median of 244 days) necessitates a need for alternative and adjunctive medications. Preclinical animal trials involving cannabidiol (CBD), one of the most prevalent cannabinoids in cannabis (marijuana) have shown its use is associated with statistically significant reductions in withdrawal symptoms and there is evidence in non-AUD populations that CBD is effective in reducing anxiety, insomnia, and seizures, which are all symptoms of alcohol withdrawal. The capacity for CBD to enhance the effect of the inhibitory neurotransmitter GABA in a manner akin to benzodiazepines has also been demonstrated. Collectively this information suggests that CBD could alleviate signs and symptoms of alcohol withdrawal, and subsequently reduce the need for adjunctive benzodiazepines.

This randomized placebo-controlled clinical trial will enroll adults with moderate-to-severe AUD who will be admitted to an inpatient research unit at the Johns Hopkins Hospital for management of their alcohol withdrawal. Enrolled participants with a history of alcohol withdrawal symptoms will be randomized to receive an oral formulation of either placebo or one of two CBD doses (10 mg/kg or 20 mg/kg). These doses have been well-studied and tolerated in prior studies and clinical trials for other disorders. Alcohol withdrawal symptoms, as defined by Diagnostic and Statistical Manual (DSM-5) criteria, will be assessed by nursing administration of the Clinical Institute Withdrawal Assessment for Alcohol, revised (CIWA-Ar) and participant completion of the Alcohol Withdrawal Symptom Checklist (AWSC). The CIWA-Ar scale will be used to guide the administration of symptom-triggered lorazepam (trade name Ativan) for all participants. As insomnia is a DSM-5 criterion for alcohol withdrawal, sleep quality will be assessed by completion of the Consensus Sleep Diary (CSD) and wrist actigraphy. Last, since cravings correlate closely with withdrawal symptoms and CBD has been observed to reduce craving for other substances, we will explore CBD's impact on alcohol craving by having participants complete the Alcohol Urge Questionnaire throughout the study. In short, the goals of this study will be to (1) determine the effect of CBD on physiologic and subjective symptoms of alcohol withdrawal, (2) determine the capacity of CBD to improve insomnia and disordered sleep during withdrawal, and (3) determine if CBD can attenuate alcohol cravings during acute abstinence.

Results from this study can help inform the possible use of CBD as a novel adjunct treatment for alcohol withdrawal and cravings that may reduce benzodiazepine need for alcohol withdrawal treatment. If CBD is shown to be effective, this line of work also points to the potential of the endogenous cannabinoid system playing a mechanistic role in alcohol's withdrawal symptoms. Finally, this study could provide further insights into the efficacy of CBD as a sleep agent for participants with alcohol withdrawal and lay the groundwork for subsequent studies exploring CBD's use in the treatment of alcohol withdrawal in an outpatient setting.

ELIGIBILITY:
Inclusion Criteria

* Meets DSM-5 criteria Moderate or Severe Alcohol Use Disorder
* Age 21-65
* Report at least one prior episode of alcohol withdrawal symptoms at least one day in duration that caused significant impairment in functioning (i.e., unable to attend work or engage in typical activities) AND/OR required medications to manage symptoms.
* Drinking at least 8 drinks a day over the two weeks prior to screening.
* Negative human chorionic gonadotropin (hCG) on qualitative urine pregnancy screen
* Shipley vocabulary score > 18, corresponding to 5th grade reading level.
* Demonstrated understanding of informed consent and ability to consent to participation in the study.

Exclusion Criteria

* Current or past alcohol-related medical complications including but not limited to cirrhosis of the liver, esophageal varices, pancreatitis, severe gastritis, hemoptysis, hematochezia, or melena.
* Use of gabapentin, benzodiazepines, or other sedative-hypnotic medications within the week prior to admission
* Regular use (e.g., more than twice a week) of cannabis or CBD products.
* Regular use of benzodiazepines (e.g., twice a week or more) within the last three months
* Meet DSM-5 criteria for moderate-to-severe substance use disorder (SUD), including Cannabis Use Disorder (except for alcohol and tobacco)
* Urine drug screen indicating the presence of substances other than cannabis at screening.
* Unstable and/or compromising medical or psychiatric conditions that would interfere with participant safety as determined by study physician.
* Current pregnancy
* BMI <17
* History of anorexia nervosa or bulimia in the past 2 years
* History of seizures or seizure disorder outside of alcohol-withdrawal related seizures
* Systolic blood pressure (SBP) > 180, Diastolic Blood Pressure (DBP) > 120 or pulse > 120 during screening or upon admission
* Any of the following laboratory values during screening or upon admission:

  * AST > 165 U/L (normal range 19-55)
  * ALT > 216 U/L (normal range 19-72)
  * Alkaline phosphatase > 378 U/L (normal range 38-126)
  * Total bilirubin >2.5 mg/dl (normal values=0.3-1.0 mg/dL)
  * Non-fasting glucose > 250 mg/ml (normal range 65-179)
  * Hematocrit < 38 % (normal range 41-53)
  * Hemoglobin < 12 g/dl (normal range 13.5-17.5) or any other laboratory value significantly outside the normal range
* Use of a prescription medication (except for birth control prescriptions) within 14 days of study entry, which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject. This includes any medication in which CYP2C9, CYP2C19, CYP1A2, CYP2B10, or CYP3A4 enzymes are major metabolizers.
* ECG with corrected QT interval (QTC) >/= 500 ms and/or presence of clinically significant abnormality
* Participation in other clinical trials within the past 60 days
* Court-mandated participation in alcohol treatment or pending incarceration

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Peak score on the Alcohol Withdrawal Symptom Checklist (AWSC) | Four times daily during inpatient stay (4 nights)
  The Alcohol Withdrawal Symptom Checklist (AWSC) is a validated measure in which participants report their own withdrawal symptoms. The scale consists of 17 items. The total possible score is 0-68, with higher scores indicating more severe withdrawal symptoms. The highest score for a participant across the duration of their time on the Clinical Research Unit (CRU) will be included in the analysis.
Peak score on the Clinical Institute Withdrawal Assessment for Alcohol, revised (CIWA-Ar) | 4 times daily during inpatient stay (4 nights)
  The Clinical Institute Withdrawal Assessment for Alcohol, revised (CIWA-Ar) is a clinically administered measurement that represents the gold standard for assessing the severity of withdrawal symptoms. It consists of 10-items: nausea/ vomiting, tremor, paroxysmal sweats, anxiety, agitation, tactile disturbances, auditory disturbances, visual disturbances, headache, and orientation/clouding of sensorium. Each sign and symptom is rated on a Likert scale from 0-7 (with 0=absent and 7 =most severe), except for "clouding of sensorium," which is ranked from 0 to 4. Scores on the CIWA-Ar scale range from 0 to 67, with higher scores indicating more severe withdrawal. The highest score for a participant across the duration of their time on the CRU will be included in the analysis. Clinical staff will use these scores to justify administration of benzodiazepines to treat withdrawal symptoms.
Average total sleep time (minutes) and wake after sleep onset as measured by wrist actigraphy | 4 nights during inpatient stay
  Actigraphy will provide a primary assessment of sleep outcomes including total sleep time and wake after sleep onset. The actigraphy devices used will be triaxial accelerometers from GT0X Link Wrist Actigraphy, Actigraph LLC. Values for total sleep time and wake time after sleep onset will be averaged across the study's four nights; this average will be included in the analysis.
Peak alcohol craving as measured by scores on the Alcohol Urge Questionnaire (AUQ) | Four times daily during inpatient stay (4 nights)
  The Alcohol Urge Questionnaire (AUQ) is an eight-item self-report questionnaire that has demonstrated validity and discriminative value in identifying and measuring alcohol craving. Each item is ranked on a score of 0 to 7, with a maximum score range of 0- 56. Higher scores indicate greater craving. The highest score for a participant across the duration of their time on the CRU will be included in the analysis.

SECONDARY OUTCOMES:
Average Total Sleep Time (minutes) as reported in Consensus Sleep Diary (CSD) results | Upon waking each morning during inpatient stay (4 days)
  The Consensus Sleep Diary (CSD) is a standardized subjective sleep rating measure in which participants rate features of their sleep-average total sleep time. Generally higher number is better.
Total Amount of Time (minutes) on Awakenings, as reported in Consensus Sleep Diary (CSD) results | Upon waking each morning during inpatient stay (4 days)
  The Consensus Sleep Diary (CSD) is a standardized subjective sleep rating measure in which participants rate features of their sleep- total amount of time on awakenings. Higher number indicating more awakenings (worse).
Sleep Quality as reported in Consensus Sleep Diary (CSD) results | Upon waking each morning during inpatient stay (4 days)
  The Consensus Sleep Diary (CSD) is a standardized subjective sleep rating measure consisting of nine items in which participants rate features of their sleep--sleep quality either "Very Poor," "Poor," "Fair," "Good," or "Very Good"
Sleep Latency (minutes) as reported in Consensus Sleep Diary (CSD) results | Upon waking each morning during inpatient stay (4 days)
  The Consensus Sleep Diary (CSD) is a standardized subjective sleep rating measure consisting of nine items in which participants rate features of their sleep - sleep latency (how long it takes one to fall asleep). Higher values would indicate worse sleep latency.
Number of Awakenings as reported in Consensus Sleep Diary (CSD) results | Upon waking each morning during inpatient stay (4 days)
  The Consensus Sleep Diary (CSD) is a standardized subjective sleep rating measure consisting of nine items in which participants rate features of their sleep--number of awakenings. Higher number indicating more awakenings (worse).
Total amount of time (minutes) spent awake after sleep onset as reported in Consensus Sleep Diary (CSD) results | Upon waking each morning during inpatient stay (4 days)
  The Consensus Sleep Diary (CSD) is a standardized subjective sleep rating measure consisting of nine items in which participants rate features of their sleep-- total amount of time spent awake after sleep onset. higher values indicating more time awake (worse).
Total doses of lorazepam administered | Every 4 hours during inpatient stay (4 nights)
  Lorazepam (trade name: Ativan) is a benzodiazepine that is frequently used in clinical practice to manage alcohol withdrawal symptoms. Since the decision to administer lorazepam is guided by CIWA scores, it can serve as a proxy for severity of withdrawal symptoms. Every four hours daily as needed for CIWA scores >/=10 while the participant stays on the inpatient Johns Hopkins Hospital (JHH) CRU
Serum levels of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) | Morning prior to admission, morning of discharge (day 5)
  Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are enzymes that act as proxies for hepatic function and damage. Elevations in the serum levels (U/L) of these enzymes--particular at levels >/= 3 times the upper limit of normal--can indicate liver injury.

CONTACTS AND LOCATIONS:
Overall Officials: David Woliinsky, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No